CLINICAL TRIAL: NCT02771821
Title: Promoting Healthy Habits With Elderlies Diabetics: Evaluation of Operative Groups as Therapeutic Intervention
Brief Title: Promoting Healthy Habits With Elderlies Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Anna Karla de Oliveira Tito Borba, Master, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAEE - 123965413.0.0000.5208
Record Dates: First submitted 2016-05-07; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus, Type 2; Aged; Health Behavior; Group Processes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Intervention (Experimental): Individual routine consultation with the Family Health Unit team and participation in operative groups based on methodology of problematization
  Interventions: Other: Operative groups based on methodology of problematization
- Control Group (No Intervention): Individual routine consultation with the Family Health Unit team

INTERVENTIONS:
Other: Operative groups based on methodology of problematization — The educational intervention based on the methodology of problematization consisted of the survey prior knowledge on the subject; planning; Implementation and Evaluation through verbalization solutions applicable to the reality of the elderlies.
  Each operative group was composed of an average of 12 to 15 elderlies diabetics who participated in monthly activities lasting 2 hours, for six consecutive months.
  Arms: Group Intervention

SUMMARY:
Randomized clinical trial with the objective of evaluating the effectiveness of operative groups to promote healthy habits in elderlies diabetics. The study was conducted in the Family Health Units of Microregion 4.2 Sanitary District IV of Recife, Pernambuco, Northeast Brazil. Participated in 202 elderlies diabetic randomly assigned to two groups: intervention and control, with similar characteristics in relation to age. Data collection occurred from August 2014 to August 2015 and elderlies were followed for 6 months (T0 to T6). Control group participated in the routine individual consultation with the staff of the Family Health Unit on a quarterly basis. Intervention group participated the routine individual consultation with the staff of the Family Health Unit on a quarterly basi and six operative groups of health education, with monthly frequency and duration of two hours, using the methodology of problematization (FREIRE, 2011), with themes identified from the needs of the participants.

DETAILED DESCRIPTION:
The study was conducted in the Family Health Units Microregion 4.2, Sanitary District IV, located in the city of Recife, Northeast Brazil. For the sample size was considered alpha error 5% (u), beta error of 20% (v). The standard deviation of glycated hemoglobin concentration distribution in both groups (Dp1 and Dp2) was equal to 1.9g/dL, and the difference between the intergroup glycated hemoglobin average was equal to 0.8%.

Initially a survey was conducted of elderlies diabetics interested in participating in the study. Then, an individual randomization of the sample was done using a table of random numbers generated by the software EPI INFO, version 6.04d. Two groups were formed, intervention and control, with similar characteristics in terms of age. Data collection occurred from August 2014 to August 2015 and the elderlies participants in the intervention group or control were followed for 6 months (T0 to T6).

Control Group: 101 elderlies diabetics who participated in the routine individual consultation with the staff of the Family Health Unit on a quarterly basis.

Group Intervention: 101 elderlies diabetics that in addition to individual routine consultation with the staff of the Family Health Unit on a quarterly basis participated in operative groups of health education. The groups had monthly frequency, duration of two hours and were conducted in close community spaces Health Units to facilitate the access of the elderlies.The operative groups with the methodology of problematization (FREIRE, 2011), included issues related to the promotion of healthy habits, identified from the needs of elderlies themselves.

In both groups, intervention and control the variables investigated were:

sociodemographic (T0) - Baseline; Knowledge about diabetes (T0 and T6) assessed by the Diabetes Knowledge Scale (DKN-A); Attitude for self-care (T0 and T6) measured by the ATT-19 - Baseline and Follow-up; healthy food consumption (T0 and T6) assessed by the Healthy Eating Index (HEI) - Baseline and Follow-up; Physical activity (T0 and T6) measured by the International Physical Activity Questionnaire (IPAQ) - Baseline and Follow-up; Anthropometric (T0 to T6) by weight measurement, height, waist circumference and body mass index - Baseline three months and follow-up; Biochemical assessment (T0, T3 and T6) by measuring glycated hemoglobin (A1C) - baseline, three months and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Elderlies people with diabetes mellitus diagnosis recorded in the medical record in the Family Health Units, located in the city of Recife, Northeast Brazil

Exclusion Criteria:

* Live in long-stay institutions
* Elderly hospitalized
* Wheelchair users
* Deficit communication and / or cognition recorded in the chart
* Presence of chronic complications of diabetes in advanced stages
* Locomotion difficulty restricting access to health facility

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Diabetes Knowledge | Six months
  Minimum score of 8 points in Diabetes Knowledge Scale (DKN-A) between the baseline and 6 months
Attitude for self-care in diabetes | Six months
  Count minimum of 70 points in the attitude questionnaire about diabetes (ATT-19) between the baseline and 6 months
Healthy food consumption | Six months
  Score larger 100 points indicating a feeding good quality through the Healthy Eating Index between the baseline and 6 months
Physical Activity | Six months
  Greater physical activity than 150 min/week in the International Physical Activity Questionnaire (IPAQ) between the baseline and 6 months
Glycated Hemoglobin | Six months
  Decrease in glycated hemoglobin levels verified by blood dosage based in change of at least 0.8% between the baseline and 6 months

SECONDARY OUTCOMES:
Body mass index | Six months
  Reduction of body mass index between the baseline and 6 months
Waist Circumference | Six months
  Reduction of waist circumference between the baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Freire P. Educação como prática de liberdade. 34ª ed. Rio de Janeiro: Paz e Terra; 2011